CLINICAL TRIAL: NCT06572046
Title: STOP-HSP.Net: a Registry for Hereditary Spastic Paraplegia as an Integration Tool for Future Therapeutic Strategies
Status: Recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: IRCCS Eugenio Medea (Other); Università degli studi di Messina (Unknown); IRCCS Istituto delle Scienze Neurologiche di Bologna (Other); Catholic University of the Sacred Heart (Other); CINECA (Unknown); Fondazione Telethon (Other)
Responsible Party: Principal Investigator, Filippo Maria Santorelli, Director of Molecular Medicine, IRCCS Fondazione Stella Maris
Other Study IDs: STOP-HSP.net
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hereditary Spastic Paraplegia
MeSH Terms: conditions — Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Blood, urine, skin biopsy, muscle biopsy, cerebrospinal fluid (all samples are optional)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our goal is to create a solid and harmonious disease registry of patient affected by hereditary spastic paraplegia (HSP) that facilitates the collection and management of patients' data over time encouraging the research and the development of future clinical trials. In-depth clinical phenotyping will develop significant clinical outcome measures that can be used in clinical trials and will allow the phenotypic complexity of the disease to be captured with the use of validated clinical scales, biomarkers and so-called patient reported outcomes (PROs).

DETAILED DESCRIPTION:
The registry will involve five recruiting clinical centres (IRCCS Fondazione Stella Maris in Pisa, IRCCS Eugenio Medea in Conegliano, IRCCS Policlinico Gemelli in Rome, IRCCS Istituto di Scienze Neurologiche in Bologna, Università degli studi di Messina) and a data analysis partner (CINECA).

Participants will be assessed annually at one of the five participating clinical sites. For each patient, at least one follow-up visit will be scheduled at an interval of 12 months in order to monitor and compare the longitudinal progression of HSP in similar groups (for example based on phenotype, age at onset, or genotype). At each visit all enrolled subjects will carry out a clinical-instrumental evaluation as per clinical practice, including: anamnestic collection, general and neurological objective examination; administration of illness scales (e.g. the SPRS scale) and quality of life questionnaires. Any biological samples will be collected as tissues, blood or urine and stored in the laboratories or bio-repositories of the individual centers and also reported in the electronic clinical report form (CRF) of STOP-HSP.net. The results of further diagnostic tests carried out such as Optical coherence tomography (OCT), brain magnetic resonance imaging (MRI) or neurophysiology performed during diagnostic practice or clinical follow up will also be collected. Any further clinical scales/evaluation questionnaires to be administered will be selected according to clinical need based on the neurological characteristics and genotype of each participant. All data relating to further instrumental and/or neurophysiological investigations carried out by the patient for clinical needs will also be collected.

The data collected during the aforementioned clinical-instrumental-laboratory evaluations will be entered into the STOP-HSP.net register in pseudonymized form.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of pure or complex HSP/spastic ataxia, even in the absence of a known genetic diagnosis
* participants/parents/legal guardians will have to give informed consent for enrollment in the registry and privacy data management

Exclusion Criteria:

* subjects affected by secondary forms of HSP
* presenting comorbidities that affect the general clinical picture according to clinical judgment
* lack of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects affected by HSP both with a known genetic diagnosis and in the absence of genotypic characterization
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishment of the STOP-HSP.net disease registry to systematically document the clinical presentation and natural history of patients affected by both pediatric-onset and adult-onset HSP | five years
Definition of genotype-specific disease progression measured by evaluating the scores of the clinical scale "Spastic Paraplegia Rating Scale" (SPRS) | five years
  Spastic Paraplegia Rating Scale (SPRS) is a 13-item scale designed to rate motor impairment in pure or complex forms of spastic paraplegia. Its score varies from 0 to 52, whereas higher scores indicate greater motor impairment.
Identification of new genetic forms of HSP through the use of Whole Genome Sequencing (WGS) in selected familial cases | five years

CONTACTS AND LOCATIONS:
Overall Officials: Filippo M Santorelli, Dr., Principal Investigator — IRCCS Fondazione Stella Maris
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data collected during the clinical-instrumental-laboratory evaluations will be entered into the STOP-HSP.net register in pseudonymized form. Each patient will be identified by a progressive code of the electronic CRF together with a unique alphanumeric identification code (automatically generated). This identification code will be used by the Center in place of the relevant name in each communication of the linked data. The Recruiting Center will be the only and exclusive entity able to associate the identification code with the personal data. The data collected in the STOP-HSP.net register will be stored on the Cloud HPC virtual infrastructure provided by CINECA on Italian territory in pseudonymized form.
Supporting Information: Study Protocol, SAP, CSR